CLINICAL TRIAL: NCT05680909
Title: Evaluation of SaCo Videolaryngeal Mask Airway for Airway Management and Intubation in Morbidly Obese Anesthetized for Elective Surgery.
Brief Title: Evaluation of SaCo Videolaryngeal Mask Airway in Morbidly Obese
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Medical University of Lodz (Other)
Responsible Party: Sponsor
Other Study IDs: RNN/104/22/KB
Record Dates: First submitted 2022-07-18; First posted 2023-01-11 (Actual); Last update posted 2023-01-11 (Actual); Status verified 2023-01

CONDITIONS: Morbid Obesity; Airway Complication of Anesthesia; Intubation Complication; Intubation; Difficult or Failed
Keywords: morbid obesity; endotracheal intubation; laryngeal mask airway; airway management
MeSH Terms: conditions — Obesity, Morbid

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- SaCo VLM evaluation: Prospective group of morbidly obese patients scheduled for elective bariatric procedure with the use of SaCo VLM for airway management.
  The following features related to SoCo VLM use will be recorded: insertion of SaCo VLM, evaluation of ventilation parameters, attempt of endotracheal intubation via SaCo VLM's lumen under continuouis visualisation of entrance to larynx using videoscope intergatred system

SUMMARY:
SaCo videolaryngeal mask airway is a novel third generation supraglottic device allowing for continuous observation of entrance to larynx via inserted in special channel videoscope connected with cable with external monitor. In obese patients airway management can be difficult so use of new devices that improve safety and potentially efficacy of airway management is indicated. In prospective observational study the SaCo VLM will be evaluated in terms of maintaining airway patency and effectiveness of intubation through it's lumen in morbidly obese scheduled for elective general surgery under general anesthesia.

DETAILED DESCRIPTION:
Morbidly obese patients pose challenge to operator when airway management is needed. Additionally they are at increased risk of complications related to failed airway management, hypoxia and following brain injury. SaCo videolaryngeal mask airway is a nowvel third generation supraglottic device allowing for continuous observation of entrance to larynx via inserted in special channel videoscope connected with cable with external monitor. In obese patients airway management can be difficult so use of new devices that improve safety and potentially efficacy of airway management is indicated.

In prospective observational study the SaCo VLM will be evaluated in terms of maintaining airway patency and effectiveness of intubation through it's lumen in morbidly obese scheduled for elective general surgery under general anesthesia.

After induction to general anesthesia SaCo VLM will be inserted with continuous visualisation through camera channel and inserted videoscope and mechanical ventilation will be commenced. Ease of SaCo VLM insertion will be recorded in 5 grade scale: 1- very easy, 2- easy, 3- neutral, 4 - difficult, 5 - very difficult. Time of insertion will be recorded as time from grabbing device and opening of patient's mouth to connecting SaCo VLM to ventilator and confirming of patient's ventilation. Parameters of mechanical ventilation will be recorded: Peak pressure, Lung Compliance - from respirator monitoring system and Seal pressure (measured with following method: fresh gas flow 5 l/min, valve set at 40cmH2O, manual/spontaneuous ventilation mode - with increasing airway pressure when the leak will be recognized achieved maximum pressure will be recorded). The visualisation of entrance to larynx will be assessed on device's monitor in 4-grade scale: 1- best view - all structures of vocal cords visible, 2 - vocal cords partialy visible, 3 - only lower part of entrance to larynx visible, 4 - no visualisation of entrance to larynx). Necessary adjustements will be reorded like external pressure on thyroid cartilage, changing of SaCo VLM mask position. In case of not adequate ventilation following steps will be taken: reposition of SaCo VLM, changing of size of SaCo VLM, endotracheal intubation using videolaryngoscope. After measurements the endotracheal intubation efforts will be commensed under continuous visualisation of entrance to larynx with SaCo VLM videoscope system. Time of intubation will be recorded. Ease of intubation will be recorded in 5 grade scale: 1- very easy, 2- easy, 3- neutral, 4 - difficult, 5 - very difficult. After successful endotracheal intubation confirmed with EtCO2 the standard general anesthesia will continue. After surgery and anesthesia the possible complications will be evaluated: track of blood on device, laryngospasm, sore throat.

ELIGIBILITY:
Inclusion Criteria:

* morbid obesity defined as BMI>40 kg/m2
* scheduled for elective surgery under general anesthesia with endotracheal intubation

Exclusion Criteria:

* lack of conscent
* airway abnormalities like for example tumors in mouth, tongue, airway injury,
* surgery on airway,
* emergency surgery,

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: morbidly obese patients scheduled for elective bariatric procedure
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-05-20 (Actual); Primary Completion 2023-01-01 (Estimated); Study Completion 2023-08-01 (Estimated)

PRIMARY OUTCOMES:
effectiveness of insertion of SaCo VLM for airway management in morbidly obese | immediate - right after performing insertion of SaCo mask
  evaluation of insertion effectiveness: proper insertion confirmend by presence of EtCO2
effectiveness of ventillation using SaCo mask in morbidly obese | immediate - right after insertion of SaCo mask
  evaluation of ventillation effectiveness indicated by proper ventilation parameters
effectiveness of visualisation of larynx using SaCo VLM in morbidly obese | immediate - right after insertion of SaCo VLM
  visualisation of entrance to larynx with intergrated SaCo VLM videoscope system - evaluated in 4 grade scale: 1 - best visualisation - all structures of entrance to larynx visible, 4 - only epiglottis visible
seal pressure of SaCo VLM in morbidly obese | immediate - right after insertion of SaCo VLM
  seal pressure - measured on anesthesia machine

SECONDARY OUTCOMES:
effectiveness of SaCo VLM for endotracheal intubation in morbidly obese | immediate - right after endotracheal intubation through SaCo mask
  evaluation of endotracheal intubation through SaCo VLM lumen: intubation confirmed by proper positioning of tube visible on monitor of device and confirmed by proper ventilation and presence of EtCO2; evaluation of easiness of ET insetion - if additional maneouvers were necessary like external pressure on thyroid cartilage.

CONTACTS AND LOCATIONS:
Overall Officials: Tomasz Gaszynski, Prof, Principal Investigator — Medical University of Lodz, Poland
Locations (1):
- Medical University of Lodz, Poland, Lodz, Poland

IPD SHARING:
Plan to Share IPD: No